CLINICAL TRIAL: NCT01003054
Title: Busulfan, Cyclophosphamide, Imatinib Mesylate and Autologous Stem Cell Transplantation in Patients With Chronic Myelogenous Leukemia
Brief Title: Autologous Transplantation for Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-672
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Leukemia; CML; Busulfan; Busulfex; Myleran; Cyclophosphamide; Cytoxan; Neosar; Imatinib Mesylate; Gleevec; Autologous Stem Cell Transplantation; Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — Busulfan; Cyclophosphamide; Imatinib Mesylate; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Transplantation (Experimental): Busulfan 130 mg/m^2 intravenous (IV) every 24 hours Days -7 to -4; Cyclophosphamide 60 mg/kg over 4 hours Day -3 and -2; Imatinib Mesylate Starting dose 100 mg/day, and Autologous Stem Cell Transplantation on Day 0.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Imatinib Mesylate; Procedure: Autologous Stem Cell Transplantation

INTERVENTIONS:
Drug: Busulfan — 130 mg/m^2 in normal saline over three (3) hours IV every twenty-four (24) hours for four (4) consecutive days (days -7 to -4)
  Other Names: Busulfex; Myleran
Drug: Cyclophosphamide — 60 mg/kg in 500 ml of normal saline over 4 hours on each of 2 consecutive days (day -3, -2)
  Other Names: Cytoxan; Neosar
Drug: Imatinib Mesylate — Starting dose 100 mg/day (mg/d), escalated to maximal dose of 400 mg/d as tolerated, after day 28 when Absolute neutrophil count (ANC) is >1500/mcl and platelets >50,000 /mcl, may be titrated to maintain ANC >1.0 and platelets >50,000 /mcl.
  Other Names: Imatinib; Gleevec; STI571; NSC-716051
Procedure: Autologous Stem Cell Transplantation — Stem Cell Infusion: Unpurged hematopoietic stem cells administered intravenously on day 0.
  Other Names: Stem Cell Transplant

SUMMARY:
The goal of this clinical research is to learn if treatment with high-dose busulfan and cyclophosphamide plus autologous bone marrow transplantation followed by treatment with Gleevec (imatinib mesylate) is effective in treating chronic myelogenous leukemia (CML).

Objectives:

1. To assess the efficacy of high dose busulfan-cyclophosphamide and autologous hematopoietic transplantation with post transplant Imatinib mesylate for the treatment of CML. The primary endpoint of the study is to determine the proportion of patients with CML alive in cytogenetic remission at one year following this treatment.
2. Secondary endpoints are time to progression and survival.

DETAILED DESCRIPTION:
Busulfan and cyclophosphamide are chemotherapy drugs which were designed to kill leukemia cells. An autologous bone marrow transplant is given after treatment with busulfan and cyclophosphamide to help in the recovery of blood and immune cells after this treatment. Imatinib mesylate is a drug which helps to stop the growth of leukemia cells. It is given after the transplant to help kill any remaining leukemia cells.

Before treatment, you will have a complete physical exam. You will have approximately 4 tablespoons of blood drawn for tests to check on the status of the disease, to check organ functions, and to check for infectious diseases (hepatitis, HIV, etc.). You will have a sample of bone marrow collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anaesthetic and a small amount of bone marrow is withdrawn through a large needle. All of these tests are being done to make sure you are eligible for this treatment. If you are found to have a "blast crisis," you will not be eligible to continue on this study.

If you are eligible or if it has not already been done recently, you will be taken to the operating room and have around 4-6 cups of bone marrow collected. The procedure will be performed under general anesthesia. The procedure is similar to the bone marrow collection at the start of the study, however, more bone marrow will be collected. The bone marrow that is collected will be frozen and stored to be given back to you after high dose chemotherapy. Before the procedure, you will be asked to donate blood (if possible). This blood will be given back to you after the procedure to replace the bone marrow that was collected. You may also need a blood transfusion from another donor.

For patients who cannot undergo the procedure of bone marrow harvesting or if not enough bone marrow was collected during the bone marrow harvesting procedure, stem cells may be collected from the blood. Normally, there are very few stem cells in the blood. Most of them are in the bone marrow. To help move or "mobilize" the cells needed from your bone marrow to your blood, you will be given injections under the skin once a day of a drug called G-CSF. The injections may given by a nurse in the hospital, in the outpatient setting, or you may learn how to give the injection yourself. Blood samples (1 tablespoon) will be drawn every day to see if there are enough stem cells in your blood. After 4-6 days of treatment with G-CSF, you will undergo a procedure called leukapheresis. This procedure is similar to donating blood to a blood bank. Blood is collected and run through a machine that processes the blood and separates the cells needed for transplantation, giving the rest back to you. The separated cells are frozen and stored to give back you after high dose chemotherapy. You may need up to 3 leukapheresis procedures to collect enough cells.

Patients who had adequate amounts of their bone marrow or blood stem cells harvested in the past will not need additional harvesting of stem cells.

At a future time when the leukemia shows signs of growth, you will have a catheter (small, flexible tube) inserted under the collar bone into a large vein in the chest. This catheter will allow the chemotherapy drugs, fluids, and other medications to be given more easily. You will have approximately 4 tablespoons of blood drawn for tests to check on the status of the disease, to check organ functions, and to check for infectious diseases (hepatitis, HIV, etc.). You will have a sample of bone marrow collected. You will also have heart (cardiac ejection fraction) and lung function tests.

You will be admitted to the hospital to receive high dose chemotherapy. You will be given busulfan by continuous injection (using the catheter) for 4 days, then you will be given cyclophosphamide by a continuous injection (using the catheter) for 2 days. The amount of busulfan you receive may be adjusted to help decrease the risk of developing side effects. You may also receive antibiotics, fluids, and other medications if your doctor feels it is necessary.

After high dose chemotherapy, you will be given your stored bone marrow or blood stem cells back ("transplant"). They will be given back to you through the catheter to help restore blood production and immunity after high dose chemotherapy. To help speed up the recovery of white blood cells, you will also be given G-CSF by injection under the skin daily until the white blood count has recovered (usually 2 to 3 weeks). You may also receive antibiotics, fluids, and other medications if your doctor feels it is necessary. Blood tests are repeated several times per week until blood counts are fully recovered and any side effects of the high dose therapy have resolved.

After your blood counts have recovered, you will begin treatment with imatinib mesylate by mouth for up to 1 year. You may also receive medications to help prevent infections for around 6 months after the transplant. These medications are usually pills to help prevent pneumonia and viral infections. While you are taking imatinib mesylate you will have blood collected (1- 4 tablespoons) for routine tests . The frequency of these blood collections will depend on your medical condition.

Around 1, 3, 6, 12, 18, and 24 months after transplant, you will have check-up visits. At these visits, you will have blood collected (1- 4 tablespoons) for routine blood tests and have a sample of bone marrow collected for tests. This bone marrow collection will be repeated 3, 4, and 5 years after the transplant procedure.

This is an investigational study. All of the drugs used in this study are FDA approved and are commercially available. Up to 50 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for hematopoietic stem cell collection and cryopreservation: a- Patients with Philadelphia chromosome positive CML < age 70 who achieve a cytogenetic remission (no Ph+ cells on bone marrow cytogenetics, at least twenty metaphases counted) are eligible for hematopoietic stem cell collection and cryopreservation. b- Patients must have a Zubrod PS <2. c.Creatinine < 1.8 mg/dl d.Serum bilirubin < 1.5 mg/dl e. SGPT < 3 x normal values f. Patients with an HLA identical sibling are eligible if they refuse allogeneic transplantation.
2. Patients are eligible for high dose therapy and autologous transplantation if they meet the following criteria (numbered 2-13): - Cytogenetic relapse characterized by > 10% Ph+ metaphases (by FISH analysis or > 2 of 20 Ph+ metaphases on 2 consecutive cytogenetic studies at least 1 month apart).
3. Cytogenetic relapse (as above) with hematologic remission or chronic phase disease, or
4. Accelerated phase or second or subsequent chronic phase.
5. Availability of stored autologous hematopoietic stem cells collected when the patient was in cytogenetic complete remission (0 of >= 20 metaphases positive for Ph+ cells).A minimum of 0.5 x 10 6 CD34 positive cells/kg or 1 x 10 8 total nucleated cells/Kg must be available.
6. Age < 70 years.
7. Zubrod PS <=2.
8. Creatinine < 1.8 mg/dL.
9. Cardiac ejection fraction > 40%.
10. DLCO > 50% of the predicted value.
11. Serum bilirubin < 1.5 mg/dL.
12. SGPT < 3 x normal values.
13. Patients with an HLA identical sibling are eligible if they refuse allogeneic transplantation.

Exclusion Criteria:

1. Uncontrolled life-threatening infections or comorbid condition that could impair tolerance to the regimen.
2. HIV positivity.
3. Pregnant or lactating women.
4. Blast crisis (>30% blasts in blood or marrow)
5. Hepatitis B or C positivity.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with CML alive in cytogenetic remission at one year following treatment | Baseline to 1 Year post treatment, up to 18 months
  Cytogenetic complete remission confirmed via bone marrow examination for morphology, cytogenetics or Fluorescence in situ hybridization (FISH).

CONTACTS AND LOCATIONS:
Overall Officials: Marcos de Lima, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org